CLINICAL TRIAL: NCT06764706
Title: A Prospective, Real-World Study EvalUating the EffectiveNess and Safety of RISankizumab in PatiEnts With Ulcerative Colitis (SUNRISE-UC)
Brief Title: Study to Assess Change in Disease Activity of Risankizumab Treatment in Adult Participants With Moderate to Severe Ulcerative Colitis
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-544
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Risankizumab; SKYRIZI
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Risankizumab: Participants will receive risankizumab as prescribed by their physician according to local label.

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine). This study will assess the change in disease activity of risankizumab treatment in adult participants with moderate to severe UC in real-world clinical practice.

Risankizumab is an approved drug for treating participants with ulcerative colitis. Approximately 200 participants who are prescribed risankizumab by their physician in accordance with local label will be enrolled in approximately multiple sites across Germany and Austria.

Participants will receive risankizumab as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 52 weeks.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with an endoscopically confirmed diagnosis of moderate to severe ulcerative colitis.
* Participants initiating risankizumab at the investigator's discretion as part of their routine clinical care; the decision to administer risankizumab must be made prior to and independent of documentation for the study and according to the approved local label.

Exclusion Criteria:

* Participants previously exposed risankizumab
* Participants who are currently participating in interventional research (not including noninterventional studies, post-marketing observational study (PMOS), or registry participation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate to severe ulcerative colitis being treated with risankizumab.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Symptomatic Remission Responder Per Partial Adapted Mayo Score | Up to approximately 52 weeks
  Symptomatic remission is defined as stool frequency (SFS) <=1 and rectal bleeding subscore (RBS)=0

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (50):
- Germany (50):
  - Universitaetsklinikum Heidelberg /ID# 275906, Heidelberg, Baden-Wurttemberg
  - Klinikum Ernst Von Bergmann /ID# 278268, Potsdam, Brandenburg
  - Private Practice - Dr. Kempelmann /ID# 275726, Tostedt, Hamburg
  - Gastroenterologische Schwerpunktpraxis /ID# 276701, Hanover, Lower Saxony
  - Katholisches Klinikum Bochum gGmbH /ID# 279486, Bochum, North Rhine-Westphalia
  - Evangelisches Krankenhaus Kalk /ID# 276414, Cologne, North Rhine-Westphalia
  - Dres. Kamp & Partner /ID# 275904, Minden, North Rhine-Westphalia
  - Gemeinschaftspraxis Innere Medizin /ID# 280068, Witten, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Im Loehr-Center Koblenz /ID# 275943, Koblenz, Rhineland-Palatinate
  - Gastroenterologische Schwerpunkt Praxis /ID# 279856, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Private Practice - Dr. Johannes Janschek /ID# 275877, Dresden, Saxony
  - Universitaetsklinikum Leipzig /ID# 276779, Leipzig, Saxony
  - Gesellschaft für klinische Studien /ID# 275867, Leipzig, Saxony
  - Private Practice - Dr. Thomas Zeisler /ID# 277933, Halle, Saxony-Anhalt
  - Studiengesellschaft BSF Unternehmergesellschaft /ID# 275905, Halle, Saxony-Anhalt
  - Praxisgemeinschaft Jerichow Schulze /ID# 275911, Jerichow, Saxony-Anhalt
  - Private Practice - Dr. Jaqueline Schumann /ID# 276126, Teuchern, Saxony-Anhalt
  - Gemeinschaftspraxis im Medicum /ID# 275933, Altenholz, Schleswig-Holstein
  - Praxis S. Tetzlaff /ID# 275882, Buedelsdorf, Schleswig-Holstein
  - Praxis Dr. Guenther-Tritsch /ID# 275886, Geesthacht, Schleswig-Holstein
  - Private Practice - Dr. Thormann & Dr. Bethge /ID# 275931, Kiel, Schleswig-Holstein
  - Praxis fuer Gastroenterologie /ID# 275903, Lübeck, Schleswig-Holstein
  - Fek - Friedrich-Ebert-Krankenhaus Neumünster /ID# 276105, Neumünster, Schleswig-Holstein
  - Dr. Jack Peter-Stein /ID# 276815, Jena, Thuringia
  - Tumorzentrum Nordthuringen Medizinisches Versorgungszentrum /ID# 280072, Nordhausen, Thuringia
  - Praxis Heil & Mueller /ID# 275927, Andernach
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 275884, Berlin
  - Facharztpraxis fur Gastroenterologie Karlshorst /ID# 277966, Berlin
  - Gastroenterologie im Mühlenbergviertel /ID# 275883, Berlin
  - Dres. Schick/Wesenberg /ID# 275878, Berlin
  - Gastro Studien GbR /ID# 275920, Berlin
  - Drk Kliniken Berlin - Köpenick /ID# 276277, Berlin
  - Private Practice - Dr. Jeannette Schwenzer & Dr. Sven Gruengreiff /ID# 276089, Berlin
  - Praxis Dr. Soellenboehmer /ID# 276183, Berlin
  - Krankenhaus Waldfriede /ID# 275913, Berlin
  - Praxis Dr. Spitz /ID# 275912, Berlin
  - Dres. Bauer/Doerflinger /ID# 276093, Freiburg im Breisgau
  - Private Practice - Dr. Matthias Eichler /ID# 275875, Hamburg
  - Gastroenterologie Rahlstedt /ID# 276408, Hamburg
  - GSGH Gastroenterologische Studiengesellschaft Herne GbR /ID# 275874, Herne
  - Gastroenterologe am Ettlinger Tor /ID# 279854, Karlsruhe
  - Dres. Breitschwerdt/Glas/Gurtler /ID# 276057, Leipzig
  - MVZ Gastroenterologie Leverkusen /ID# 275901, Leverkusen
  - Gastropraxis Magdeburg /ID# 275885, Magdeburg
  - Bettenworth & Partner /ID# 275900, Münster
  - Pc Docs /Id# 275876, Pirmasens
  - Praxis fuer Gastroenterologie /ID# 275946, Schwerin
  - Dres. Rehbehn/Skusa /ID# 276090, Solingen
  - Private Practice - Dr. Markus Braunfels /ID# 277129, Wesseling
  - Dr. Schirin-Sokhan /ID# 276982, Würselen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-544